CLINICAL TRIAL: NCT04402203
Title: Study on Safety and Efficacy of Favipiravir (Favipira) for COVID-19 Patient in Selected Hospitals of Bangladesh
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bangladesh Medical Research Council (BMRC) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 29318042020
Record Dates: First submitted 2020-05-19; First posted 2020-05-26 (Actual); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: COVID-19; Favipiravir (Favipira)
MeSH Terms: conditions — COVID-19 | interventions — favipiravir

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled randomized control study. Randomization will be done by computerized randomization table Group A Patient (25) = Favipiravir + Standard Treatment Group B Patient (25) = Only Standard Treatment For better result sample size may be multiply on the basis of availability of COVID-19 patient in the study hospital.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Favipiravir + Standard Treatment (Experimental): Favipiravir 200 mg (Favipira) tablet will be given orally. Day 1: Tablet Favipiravir 1600 mg twice daily Days 2-Days 10: Tablet Favipiravir 600 mg twice daily.
  Interventions: Drug: Favipiravir
- Only Standard Treatment (Placebo Comparator): Standard treatment included oxygen inhalation, oral or intravenous rehydration, electrolyte correction, antipyretics, analgesics, antibiotics and antiemetic drugs & the medication any patient is on due to any concomitant diseases.
  Interventions: Drug: Only Standard Treatment

INTERVENTIONS:
Drug: Favipiravir — Favipiravir 200 mg (Favipira) tablet will be given orally. Day 1: Tablet Favipiravir 1600 mg twice daily Days 2-Days 10: Tablet Favipiravir 600 mg twice daily.
  Arms: Favipiravir + Standard Treatment
Drug: Only Standard Treatment — Standard treatment included oxygen inhalation, oral or intravenous rehydration, electrolyte correction, antipyretics, analgesics, antibiotics and antiemetic drugs & the medication any patient is on due to any concomitant diseases.
  Arms: Only Standard Treatment

SUMMARY:
A recent outbreak of coronavirus disease 2019 (COVID-19) caused by the novel coronavirus designated as severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) started in Wuhan, China, at the end of 2019. The clinical characteristics of COVID-19 include respiratory symptoms, fever, cough, dyspnea, and pneumonia. As of 25 February 2020, at least 77 785 cases and 2666 deaths had been identified across China and in other countries; in particular, 977 and 861 cases were identified in South Korea and Japan, respectively. The outbreak has already caused global alarm. On 30 January 2020, the World Health Organization (WHO) declared that the outbreak of SARS-CoV-2 constituted a Public Health Emergency of International Concern (PHEIC), and issued advice in the form of temporary recommendations under the International Health Regulations (IHR).It has been revealed that SARS-CoV-2 has a genome sequence that is 75%-80% identical to that of SARS-CoV, and has more similarities to several bat coronaviruses. SARS-CoV-2 is the seventh reported human-infecting member of the family Coronaviridae, which also includes SARS-CoV and the Middle East respiratory syndrome (MERS)-CoV. It has been identified as the causative agent of COVID-19. Both the clinical and the epidemiological features of COVID-19 patients demonstrate that SARS-CoV-2 infection can lead to intensive care unit (ICU) admission and high mortality. About 16%-21% of people with the virus in China have become severely ill, with a 2%-3% mortality rate. However, there is no specific treatment against the new virus.

Therefore, it is urgently necessary to identify effective antiviral agents to combat the disease and explore the clinical effect of antiviral drugs. One efficient approach to discover effective drugs is to test whether the existing antiviral drugs are effective in treating other related viral infections. Several drugs, such as ribavirin, interferon (IFN), Favipiravir (FPV), and Lopinavir (LPV)/ritonavir (RTV), have been used in patients with SARS or MERS, although the efficacy of some drugs remains controversial. It has recently been demonstrated that, as a prodrug, Favipiravir (half maximal effective concentration (EC50) = 61.88 μmol·L-1, half-maximal cytotoxic concentration (CC50) > 400 μmol·L-1, selectivity index (SI) > 6.46) effectively inhibits the SARS-CoV-2 infection in Vero E6 cells (ATCC-1586). Furthermore, other reports show that FPV is effective in protecting mice against Ebola virus challenge, although its EC50 value in Vero E6 cells was as high as 67 μmol·L-1. Therefore, clinical studies are urgently needed to evaluate the efficacy and safety of this antiviral nucleoside for COVID-19 treatment. After enrollment of the patients (day 1) depending on inclusion and exclusion criteria and laboratory findings confirming the presence of the COVID-19 virus, 25 patients will receive Favipiravir plus standard treatment and the second group of 25 patients will receive standard treatment only. The comparison of the findings of the follow up studies on days 4, 7, and 10 in terms of clinical manifestations, chest X-ray and laboratory findings, such as Real Time Polymerase Chain Reaction (RT-PCR) results for viral presence will determine whether Favipiravir has safety and efficacy against COVID-19 infections.

All ethical issues related to this trial including right of the participants to withdraw from the study should be maintained according to of guidelines of International Conference on Harmonisation (ICH)-Good Clinical Practice (GCP).

DETAILED DESCRIPTION:
•Rationale: Coronavirus disease 2019 (COVID-19) is defined as illness caused by a novel coronavirus now called severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2; formerly called 2019-nCoV), which was first identified amid an outbreak of respiratory illness cases in Wuhan City, Hubei Province, China. It was initially reported to the World Health Organization (WHO) on December 31, 2019. On January 30, 2020, the WHO declared the COVID-19 outbreak a global health emergency. On March 11, 2020, the WHO declared COVID-19 a global pandemic, its first such designation since declaring influenza A virus subtype (H1N1) influenza a pandemic in 2009. No drugs or biologics have been proven to be effective for the prevention or treatment of COVID-19. Numerous antiviral agents, immunotherapies, and vaccines are being investigated and developed as potential therapies Fujifilm Toyama Chemical has started a Phase III clinical trial of its antiviral influenza drug Avigan (favipiravir) for the treatment of Covid-19 patients in Japan. Avigan specifically blocks RNA polymerase associated with influenza viral replication. The mechanism is expected to have an antiviral effect on SARS-CoV-2, the novel coronavirus that causes Covid-19. In Japan, the new Phase III trial will assess Avigan's safety and efficacy as a potential Covid-19 treatment. Last month, China's Science and Technology Ministry official Zhang Xinmin said that favipiravir helped patients recover in an 80-day participant trial conducted in Shenzhen city.

According to the study data, the drug was able to shorten the recovery time from 11 days to four days for mild and moderate cases. Favipiravir secured Chinese approval for manufacturing by Zhejiang Hisun Pharmaceutical to treat adults with new or recurring influenza. It also holds approval in China as an investigational treatment for Covid-19. A drug developed by Fujifilm Toyama Chemical in Japan is showing promising outcomes in treating at least mild to moderate cases of COVID-19, Live Science previously reported. The antiviral drug, called Favipiravir or Avigan, has been used in Japan to treat influenza, and last month, the drug was approved as an experimental treatment for COVID-19 infection. The drug, which works by preventing certain viruses from replicating, seemed to shorten the duration of the virus as well as improve lung conditions (as seen in X-rays) in tested patients.

A few studies have been published in international journals regarding the efficacy and safety of Favipiravir. However, this type of study on Favipiravir (Favipira) has not yet been done in our country. This is the rationale why we have designed this clinical trial in Bangladesh to fight against COVID-19 a global pandemic.

Objectives:

•General Objectives:

To evaluate the efficacy and safety of Favipiravir (Favipira) for the treatment of COVID-19 in a group of Bangladeshi patients

Specific objectives:

Primary end point:

•To assess the treatment efficacy: Negative for the virus at 4-10 days after initiation of therapy. However, negative results for the viral presence should be with an interval of at least 24 hours.

* To assess the treatment efficacy: X-ray findings of lung condition improvement at Day-4, Day-7 and Day-10 of therapy.

Secondary end point:

* Clinical recovery rate at 7-10 days of therapy and reduced duration of fever, cough, relief time auxiliary oxygen therapy or noninvasive mechanical ventilation rate.
* To assess the adverse effects of drug.
* ICU admission rate
* Mortality rate

Hypothesis

Favipiravir might be an effective drug for the treatment of COVID-19.

Methodology:

Study design: Double-blind, placebo-controlled randomized control study. Randomization will be done by computerized randomization table.

Place of study: Mahanagar General Hospital, Dhaka (Site-1), Mugda Medical College Hospital, Dhaka (Site-2), Kurmitola General Hospital, Dhaka (Site-3), Dhaka Medical College Hospital, Dhaka (Site-4)

Duration of study: 2 months

Study population: Clinically and Laboratory-confirmed patients with COVID-19

Formulae:

Variable Notations:

Α, the probability of type I error (significance level) is the probability of rejecting the true null hypothesis (0.05) Β, the probability of type II error (1 - power of the test) is the probability of failing to reject the false null hypothesis (0.80).

PA (proportion of discordant pairs of type A) among discordant pairs (1/4) PD (proportion of discordant) pairs among all pairs (0.25) Npairs, required sample size pair =25*2=50 A matched-pair design is used, in which patients are matched on age and clinical stage of COVID-19, with one patient in a matched pair assigned to treatment case and the other to treatment control. It is estimated that patients in a matched pair will respond similarly to the treatments in 85% of matched pairs. How many matched pairs need to be enrolled in the study to have a 90% chance of finding a significant difference using a two-sided test with type I error = 0.05? So, we will recruit a total of 50 patients

Randomization will be done by computerized randomization table Group A Patient (25) = Favipiravir + Standard Treatment Group B Patient (25) = Only Standard Treatment For better result sample size may be multiply on the basis of availability of COVID-19 patient in the study hospital.

Diagnostic Criteria

All patients diagnosed as COVID-19 positive on the basis of clinical and Laboratory findings. If the respiratory specimens give positive results upon RT-PCR analysis at the lab targeting conserved viral gene(s), such as E gene and or RNA-dependent RNA polymerase (RdRp) gene or other COVID-19 specific genes, it will be considered as confirmed positive case for COVID-19.

Data Collection Procedure:

Patient admitted in Isolation ward with COVID-19 positive will be used. Study population again will be confirmed by laboratory findings. Patients will be selected for the study following inclusion and exclusion criteria. Written consent will be taken from the patient for treatment with Favipiravir. After data collection, data will be analyzed for result. Finally, Summary and conclusion will be published.

Background of Data Collectors at the clinical sites:

Data will be collected by Co-investigators of the study who are employed as physicians in the Isolation word for COVID-19 positive patients in the designated hospitals. Co-investigators are familiar about the data collection procedure as per clinical trial protocol.

Precaution and safety of the Data Collectors including physicians, laboratory personnel, nurses, and medical technologists:

Data Collectors should fill up data collection sheet properly. Proper monitoring of the patient should be carefully done.

Data collectors must wear appropriate personal protective equipment (PPE) including gown, N95 mask, hand gloves, head coverings and goggles to protect themselves. I case, anyone involved in the study get infected, he/she should be sent to the designated isolation unit/quarantine to mitigate spread of the disease and get treatment.

Treatment:

Favipiravir 200 mg (Favipira) tablet will be given orally. Day 1: Tablet Favipiravir 1600 mg twice daily Days 2-Days 10: Tablet Favipiravir 600 mg twice daily. Group A Patient (25) = Favipiravir + Standard Treatment Group B Patient (25) = Only Standard Treatment

Standard treatment included oxygen inhalation, oral or intravenous rehydration, electrolyte correction, antipyretics, analgesics, antibiotics and antiemetic drugs & the medication any patient is on due to any concomitant diseases.

Management of adverse events:

It has been suggested that host cell enzymes (cellular kinases) convert Favipiravir into Favipiravir ribofuranosyl phosphate, a form that inhibits virus polymerase without affecting host cellular RNA or DNA synthesis. Research documents indicate that Favipiravir is a well-tolerated drug with some side effects like headache, nausea and hypersensivity. On prolong treatment it may develop inflammation of liver and kidney, abortion, intrauterine fetal death, and congenital anomalies of newborn baby.

Considering the longterm effects of Favipiravir, patients with Chronic liver and kidney disease, previous history of allergic reactions to Favipiravir, Pregnant or lactating women, Women of a childbearing age with a positive pregnancy test and having history of Miscarriage, or within 2 weeks after delivery have been excluded in the study proposal.

Management of side effects like headache, nausea and hypersensitivity will counter at the early stage of onset and all medicines and instruments will be kept available at the ward near the patient bed for prompt management during treatment with Favipiravir.

Any adverse or side effect will be managed immediately with standard treatment procedure with discontinuation of the test drug Research physicians under the supervision of Clinical Trial Monitors will monitor clinically all the vital signs along with adverse symptoms (if any arise) routinely and be available for taking measures against any side or adverse effect. They will record all the events clinically along with the routine data collection.

For any occurrence due mismanagement with the side effects of Favipiravir, the entire research team will be responsible.

Adverse Drug Reaction Reporting time:

If any adverse drug reaction occurs during study period it should be reported within 24 hours of the event to the Data Safety and Monitoring Board (DSMB) in order to assess the risk and quick action should be taken.

Laboratory data collection Blood and respiratory samples will be collected by trained medical technologist and transported immediately to Institute for developing Science and Health initiatives (ideSHi) for analysis. Cool chain will be maintained during sample transportation. Blood sample analysis at the laboratory will be done by trained research officers and fellows. On the other hand, RT-PCR using respiratory samples for viral detection will be done by expert molecular biologist.

Follow-up System:

Baseline clinical symptoms and Laboratory findings will be monitored from first day and follow up will be continued at Day-4, Day-7 and Day-10. Viral clearance will be checked by RT-PCR at Day-4, Day-7 and Day-10. X-ray findings will be monitored from Day-1 followed by Day-4, Day-7 and Day-10 to see the lung condition. Any Side effects of drugs will be documented.

Statistical Analysis:

All data will be analyzed by using the statistical package for social science (SPSS) 22. All data will be provided as mean ± standard deviation (SD). Chi-square test will be used to compare differences between the frequencies. Serum cytokines levels will be analyzed using the normality test. P value < 0.05 will be considered significant.

•Utilization of Results:

A recent outbreak of coronavirus disease 2019 (COVID-19) caused by the novel coronavirus designated as severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) started in Wuhan, China, at the end of 2019. The clinical characteristics of COVID-19 include respiratory symptoms, fever, cough, dyspnea, and pneumonia. According to world health organization (WHO), COVID-19 updates on 10th April, 2020, globally confirmed cases were 16,17,204, confirmed deaths were 97,039, recovered 364686 peoples. In Bangladesh confirmed cases were 424, confirmed deaths were 27, recovered 33 peoples.

No drugs or biologics have been proven to be effective for the prevention or treatment of COVID-19. Numerous antiviral agents, immunotherapies, and vaccines are being investigated and developed as potential therapies. A drug developed by Fujifilm Toyama Chemical in Japan is showing promising outcomes in treating at least mild to moderate cases of COVID-19, Live Science previously reported. The antiviral drug, called Favipiravir or Avigan, has been used in Japan to treat influenza, and last month, the drug was approved as an experimental treatment for COVID-19 infection. The drug, which works by preventing certain viruses from replicating, seemed to shorten the duration of the virus as well as improve lung conditions (as seen in X-rays) in tested patients.In our study on Favipiravir (Favipira), if we will get promising result regarding efficacy and safety, then it saves thousands life of Bangladeshi people. We may also export the Medicine across the globe to fight against COVID-19 a global pandemic.

* Facilities: Kurmitola General Hospital and Kuwait Bangladesh Maitry Govt. Hospital, both Hospitals are Bangladesh Govt. approved hospital for COVID-19 treatment. So, almost all facilities will be available.
* Ethical Implications:
* Permission will be taken from Bangladesh Medical Research Council and The Directorate General of Drug Administration (DGDA) for conducting this study.
* Before data collection objective of the study will be informed to the respondent.
* Informed written consent will be obtained from the participants of the study
* The privacy and confidentiality will strictly be maintained during data collection
* Right to discontinue from the study at any time will be ensured
* Any adverse or side effect will be managed immediately with standard treatment procedure with discontinuation of the test drug

ELIGIBILITY:
Inclusion Criteria:

1. Age: Male or female patients 18 -65 years old
2. Respiratory samples tested positive for the novel coronavirus.
3. Initial symptoms will within 7 days
4. Nonpregnant women (confirmed by urine human chorionic gonadotropin (HCG) test prior to enrollment)

Exclusion Criteria:

1. Severe clinical condition (meeting one of the following criteria: a resting respiratory rate greater than 30 per minute, oxygen saturation below 93%, oxygenation index (OI) < 300 mmHg (1 mmHg = 133.3 Pa), respiratory failure, shock, and/or combined failure of other organs that required ICU monitoring and treatment).
2. Chronic liver and kidney disease and reaching end stage. (Serum aspartate aminotransferase (AST) and Serum alanine aminotransferase (ALT) will be elevated over 5 times of normal upper range will excluded).

   (Normal upper limit of Serum AST = 40 units /L, ALT = 56 units /L)
3. Serum uric acid >7.0 mg/dL in Male and Serum uric acid >6.0 mg/dL in Female will excluded
4. ICU patient
5. Previous history of allergic reactions to Favipiravir.
6. Pregnant or lactating women
7. Women of a childbearing age with a positive pregnancy test.
8. Miscarriage, or within 2 weeks after delivery
9. Hypertensive patients, who are taking Calcium Channel Blockers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-05 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Number of participants negative by RT-PCR for the virus at 4-10 days after initiation of therapy. | at 4 to 10 days of therapy
  Negative by RT-PCR for the virus at 4-10 days after initiation of therapy. However, negative results for the viral presence should be with an interval of at least 24 hours.
Number of participants with lung condition change assessed with X-ray. | at Day-4, Day-7 and Day-10 of therapy
  X-ray findings of lung condition improvement at Day-4, Day-7 and Day-10 of therapy

SECONDARY OUTCOMES:
Number of participants with clinical recovery | at Day-4, Day-7 and Day-10 of therapy
  Clinical recovery indicates reduced duration of fever, cough, relief time auxiliary oxygen therapy or noninvasive mechanical ventilation rate.
Number of participants with adverse effects of drug. | at Day-4, Day-7 and Day-10 of therapy
Number of participants requiring ICU admission | at Day-4, Day-7 and Day-10 of therapy
Number of death | at Day-4, Day-7 and Day-10 of therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Mahanagar General Hospital, Dhaka (Site-1), Mugda Medical College Hospital, Dhaka (Site-2), Kurmitola General Hospital, Dhaka (Site-3), Dhaka Medical College Hospital, Dhaka (Site-4), Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Li Q, Guan X, Wu P, Wang X, Zhou L, Tong Y, Ren R, Leung KSM, Lau EHY, Wong JY, Xing X, Xiang N, Wu Y, Li C, Chen Q, Li D, Liu T, Zhao J, Liu M, Tu W, Chen C, Jin L, Yang R, Wang Q, Zhou S, Wang R, Liu H, Luo Y, Liu Y, Shao G, Li H, Tao Z, Yang Y, Deng Z, Liu B, Ma Z, Zhang Y, Shi G, Lam TTY, Wu JT, Gao GF, Cowling BJ, Yang B, Leung GM, Feng Z. Early Transmission Dynamics in Wuhan, China, of Novel Coronavirus-Infected Pneumonia. N Engl J Med. 2020 Mar 26;382(13):1199-1207. doi: 10.1056/NEJMoa2001316. Epub 2020 Jan 29. PMID 31995857
- [Background] Chen N, Zhou M, Dong X, Qu J, Gong F, Han Y, Qiu Y, Wang J, Liu Y, Wei Y, Xia J, Yu T, Zhang X, Zhang L. Epidemiological and clinical characteristics of 99 cases of 2019 novel coronavirus pneumonia in Wuhan, China: a descriptive study. Lancet. 2020 Feb 15;395(10223):507-513. doi: 10.1016/S0140-6736(20)30211-7. Epub 2020 Jan 30. PMID 32007143
- [Background] Lu R, Zhao X, Li J, Niu P, Yang B, Wu H, Wang W, Song H, Huang B, Zhu N, Bi Y, Ma X, Zhan F, Wang L, Hu T, Zhou H, Hu Z, Zhou W, Zhao L, Chen J, Meng Y, Wang J, Lin Y, Yuan J, Xie Z, Ma J, Liu WJ, Wang D, Xu W, Holmes EC, Gao GF, Wu G, Chen W, Shi W, Tan W. Genomic characterisation and epidemiology of 2019 novel coronavirus: implications for virus origins and receptor binding. Lancet. 2020 Feb 22;395(10224):565-574. doi: 10.1016/S0140-6736(20)30251-8. Epub 2020 Jan 30. PMID 32007145
- [Background] Wang M, Cao R, Zhang L, Yang X, Liu J, Xu M, Shi Z, Hu Z, Zhong W, Xiao G. Remdesivir and chloroquine effectively inhibit the recently emerged novel coronavirus (2019-nCoV) in vitro. Cell Res. 2020 Mar;30(3):269-271. doi: 10.1038/s41422-020-0282-0. Epub 2020 Feb 4. No abstract available. PMID 32020029
- [Background] Oestereich L, Ludtke A, Wurr S, Rieger T, Munoz-Fontela C, Gunther S. Successful treatment of advanced Ebola virus infection with T-705 (favipiravir) in a small animal model. Antiviral Res. 2014 May;105:17-21. doi: 10.1016/j.antiviral.2014.02.014. Epub 2014 Feb 26. PMID 24583123
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Background] Gordon CJ, Tchesnokov EP, Feng JY, Porter DP, Gotte M. The antiviral compound remdesivir potently inhibits RNA-dependent RNA polymerase from Middle East respiratory syndrome coronavirus. J Biol Chem. 2020 Apr 10;295(15):4773-4779. doi: 10.1074/jbc.AC120.013056. Epub 2020 Feb 24. PMID 32094225
- See also: Coronavirus disease 2019 (COVID-19) Situation Report — https://www.who.int/
- See also: Max Roser, Hannah Ritchie and Esteban Ortiz-Ospina — https://ourworldindata.org/coronavirus
- See also: Fujifilm commences Phase III trial of Avigan for Covid-19. — https://www.clinicaltrialsarena.com/news/fujifilm-avigan-covid-19-trial-japan/
- See also: Favipiravir (T-705), a broad spectrum inhibitor of viral RNA polymerase — https://www.jstage.jst.go.jp/article/pjab/93/7/93_PJA9307B-02/_html/-char/ja